CLINICAL TRIAL: NCT00998361
Title: Hematopoietic Stem Cell Transplantation From HLA Compatible Donor in Ewing Sarcomas and Soft Tissues Sarcomas
Brief Title: Hematopoietic Stem Cell Transplantation From Human Leukocyte Antigen (HLA) Compatible Donor in Ewing Sarcomas and Soft Tissues Sarcomas
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Collaborators: S. Anna Hospital (Other)
Responsible Party: Dr Augusto Cavina, S. Orsola-Malpighi Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CE_clin.42_2009_S_sper
Record Dates: First submitted 2009-10-18; First posted 2009-10-20 (Estimated); Last update posted 2009-10-20 (Estimated); Status verified 2009-10

CONDITIONS: Ewing; Soft Tissue Sarcoma
Keywords: Sarcoma; allogeneic; Hemopoietic stem cell transplant
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Stem Cell Transplant (Experimental): All the patient who are affected by refractory or resistant or relapsed Soft tissue sarcoma o Ewing sarcoma who find an HLA compatible allogeneic donor and are submitted to Stem cell transplantation
  Interventions: Procedure: Allogeneic hemopoietic stem cell transplant

INTERVENTIONS:
Procedure: Allogeneic hemopoietic stem cell transplant — administration of 15 mg/kg of thiotepa + 140 mg/sqm of melphalan followed by infusion of allogeneic hemopoietic stem cell
  Other Names: CE_clin.42_2009_S_sper

SUMMARY:
This is a perspective multicentric study for the treatment of patients aged equal or less than 60 years and submitted to an allogeneic hematopoietic stem cell transplantation from an HLA compatible related or unrelated donor because affected by resistent or refractory or relapsed after autologous stem cell transplantation Ewing Sarcoma or Soft tissues sarcoma who did not benefit from conventional therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age 0-60 years.
* Performance status according to Karnofsky score > 70%
* Normal liver function
* Normal renal function
* Normal cardiac function
* Informed consent
* Availability of an HLA compatible Donor

Exclusion Criteria:

* Absence of at least one of the inclusion criteria

Ages: 1 Month to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 140 (Actual)
Dates: Start 2009-06; Primary Completion 2010-06 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) a 12 months from the enrollment higher than 30% for the patients submitted to allogeneic stem cell transplantation in front of the patients who received conventional chemotherapy. | 12 months from the enrollement

SECONDARY OUTCOMES:
Transplant related mortality | 12 months after the enrollement of the first patients

CONTACTS AND LOCATIONS:
Overall Officials: Arcangelo Prete, MD, PhD, PI, Principal Investigator — S. Orsola-Malpighi Hospital
Locations (1):
- Pediatric Oncology and Hematology Department, S. Orsola-Malpighi Hospital, Bologna, Italy